CLINICAL TRIAL: NCT06034574
Title: A Trial Investigating the Accuracy of Continuous Glucose Monitor Systems ("Supersapiens" Abbott Libre Sense and Dexcom G6) During Exercise in People With Normal Glucose Tolerance
Acronym: SuperComEx
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 21HH7234
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Type 1 Diabetes
Keywords: Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Continuous glucose monitoring — Assessment of accuracy of two different continuous glucose monitoring devices during exercise

SUMMARY:
A two-phase, observational trial in an exercise laboratory and a prospective real-world setting to test the hypothesis that The Libre Sense Glucose Sport device has acceptable accuracy in people with normal glucose tolerance and comparable accuracy in the range of 3.0 to 11mmol/L to clinically approved CGM in people with type 1 diabetes.

DETAILED DESCRIPTION:
This is two-phase trial including a research facility and home phase existing of five study related visits:

* Screening visit and CPX test (2 hrs per visit)
* three exercise sessions completed in a random order at the research facility (2 hrs per visit) plus an additional visit for people with normal glucose tolerance to undertake a glucose tolerance test
* 4 weeks of home-based exercise (3 sessions of ~60 minutes moderate intensity exercise per week) - Including one glycaemic challenge prior to a single home-based exercise session
* Final visit

ELIGIBILITY:
Inclusion Criteria:

* • Male or female aged 18-65 years (both inclusive)

  * Body mass index 18.0-29.9 kg/m2 (both inclusive)
  * Normal glucose tolerance (measured via fasting blood glucose levels) or type 1 diabetes for greater than 1 year
  * Participants performing regular physical activity during the last 3 months prior to screening
  * Mass-specific peak oxygen consumption (VO2peak) >20 ml/kg/min
  * For participants with type 1 diabetes

    * Stable insulin regimen for 6 months
    * HbA1c ≤69mmol/mol

Exclusion Criteria:

* • Enrolment in other study, except at the discretion of the Chief investigator

  * Known or suspected hypersensitivity to trial product(s) or related products
  * Receipt of any investigational medicinal product within 1 week prior to screening in this trial
  * Suffer from or history of a life-threatening disease (i.e. cancer judged not to be in full remission except basal cell skin cancer or squamous cell skin cancer), or clinically severe diseases that directly influence the study results, as judged by the Investigator. This does not prohibit the participation of patients taking medications that influences the metabolism (e.g. statin) or cardio-respiratory system (e.g. asthma spray) as long as the therapy is stable and is not adapted throughout the run of the trial. Furthermore, it does not excluded patients how have celiac disease (or similar diseases or allergies), as long as the disease is stable, and patients are able to stay on their specific (e.g.) gluten-free diet.
  * Participant with a heart rate <35 beats per minute (bpm) at screening (after resting for 5 min in supine position)
  * Supine blood pressure at screening (after resting for 5 min in supine position) outside the range of 90-150 mmHg for systolic or 50-95 mmHg for diastolic (excluding white-coat hypertension; therefore, if a repeated measurement on a second screening Visit shows values within the range, the participant can be included in the trial). This exclusion criterion also pertains to participants being on anti-hypertensives
  * Significant abnormal ECG at screening, as judged by the Investigator
  * Any chronic (metabolic) disorder or severe disease which, in the opinion of the Investigator might jeopardise participant's safety or compliance with the protocol
  * History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction
  * Participant with mental incapacity or language barriers precluding adequate understanding or cooperation or who, in the opinion of their general practitioner or the Investigator, should not participate in the trial
  * Potentially non-compliant or uncooperative during the trial, as judged by the Investigator
  * Any condition that would interfere with trial participation or evaluation of results, as judged by the Investigator
  * Female of childbearing potential who is pregnant, breast-feeding or intend to become pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 16 healthy volunteers undertaking regular physical activity 8 volunteers with type 1 diabetes undertaking regular physical activity
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
%MARD lab phase | 2 weeks
  To assess % mean or median absolute relative difference (%MARD) of Supersapiens Abbott Libre Sense during exercise to reference capillary blood glucose (lab phase)

SECONDARY OUTCOMES:
%MARD home phase | 4 weeks
  To assess % mean or median absolute relative difference (%MARD) of Supersapiens Abbott Libre Sense during exercise to reference capillary blood glucose (home phase)

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Clinical Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No